CLINICAL TRIAL: NCT07227662
Title: Feasibility, Usability and Preliminary Efficacy of Home-based FES Fro Adhesive Capsulitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Kelly Westlake, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HP-00116646
Record Dates: First submitted 2025-10-27; First posted 2025-11-13 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Adhesive Capsulitis
Keywords: Functional Electrical Stimulation; Home-based; Shoulder Adhesive Capsulitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Home-based FES (Other): The intervention will include home use of Genesis Flex FES device alongside usual rehabilitation care. Participant education in Genesis FES use will be conducted during the baseline assessment session. FES parameters will be initially adjusted at the lowest possible current for patient comfort with the constraint that they should not elicit a tetanic contraction. FES will be provided via two self adhesive electrodes attached across shoulder joint.A shoulder harness adjustable neoprene padding will be provided to enable anatomical contouring for patient comfort and support for positioning of stimulator and electrodes to the affected shoulder.
  Interventions: Device: Home based FES in combination with usual therapy

INTERVENTIONS:
Device: Home based FES in combination with usual therapy — Participants diagnosed with shoulder adhesive capsulitis and being treated at a local physical and occupational therapy outpatient clinic will be deemed eligible for inclusion in the study.The intervention will include home use of Genesis Flex FES device alongside usual rehabilitation care. Usual care therapy may consist of manual therapy, hot packs, transcutaneous electrical nerve stimulation, ultrasound treatments, daily home-based shoulder exercises, and/or acetaminophen for pain, which will be documented.

SUMMARY:
The purpose of this study is to investigate the feasibility, usability and preliminary efficacy of a home-based Functional Electrical Stimulation(FES) in individuals with shoulder adhesive capsulitis. The main question it aims to answer is if combining home-based FES to usual therapy at the clinic will improve pain and improve function of the impaired shoulder.

DETAILED DESCRIPTION:
Individuals with shoulder adhesive capsulitis will be recruited. All participants will complete clinical assessments at 3 time points(baseline, 2 weeks into the intervention and 4 weeks after). Each participant will be asked to complete either one 60min or 2x30 min duration of FES daily for 4 weeks.

The following assessments will be performed:Likert rating scales and open-ended questions,The Disabilities the Arm, Shoulder, and Hand (DASH) questionnaire,Active and passive shoulder range of motion (ROM) will be assessed using goniometric measurements for shoulder flexion, abduction, and external rotation,Pain rating at rest, night, and end range movement using a visual analogue scale (0-10 points)

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Individuals diagnosed with shoulder adhesive capsulitis
3. Shoulder pain, limited shoulder mobility for more than 4 weeks, normal shoulder x-ray findings, and normal neurological exam
4. Can tolerate electrical stimulation

Exclusion Criteria:

1. Presence of shoulder tumors or bone lesions
2. History of shoulder fracture or subluxation
3. History of shoulder surgery
4. Severe osteoporosis,
5. Rheumatic disease
6. Radiating pain from cervical radiculopathy
7. Participation in other clinical trial, and/or intraarticular steroid injections within 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Participant Acceptability and Satisfaction | At the end of 4 weeks
  Participant-reported satisfaction, comfort, and ease of use assessed using a 5-point Likert scale and open-ended qualitative feedback.A Likert scale is a rating scale used in surveys to measure opinions, attitudes,and perceptions by asking respondents to indicate their level of agreement or disagreement with a statement. It consists of a series of statements with a symmetric range of response options, such as a five-point scale from 0="Strongly Disagree" to 5="Strongly Agree". This method allows for the collection of quantitative data to analyze subjective experiences.
Usability of the FES device for home-based use | At the end of 4 weeks
  Percentage of participants able to correctly and independently use the portable FES device for ≥80% of prescribed home sessions, as verified by device logs and participant self-report.

SECONDARY OUTCOMES:
Change in Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire score | Change from baseline DASH at 4 weeks
  The Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire is a 30-item self-report measure assessing symptoms and functional limitations related to upper-limb musculoskeletal disorders. It also includes two optional 4-item modules (Work and Sports/Performing Arts). Each item is rated on a 5-point scale and converted to a total score ranging from 0 to 100, where 0 indicates no disability and 100 indicates the most severe disability. Changes in DASH total and optional module scores will be compared from baseline to 4 weeks.
Change in Active and Passive Shoulder Range of Motion (ROM) | Change from baseline ROM at 4 weeks
  Active and passive shoulder ROM will be assessed using goniometric measurements for shoulder flexion, abduction, and external rotation.
Change in Shoulder Pain using Visual Analog Scale | Change from Baseline VAS at 4 weeks
  Change in shoulder pain intensity assessed using a 10-point Visual Analog Scale (VAS), where 0 = no pain and 10 = worst pain imaginable. Pain will be rated at rest, during the night, and at end-range shoulder movement.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rehman ZI, Khan S, Abbas M. Effect of FES with and without Mulligan's technique in adhesive capsulitis. J Health Rehabil Res. 2024;4(3):Article 1408
- [Background] Challoumas D, Biddle M, McLean M, Millar NL. Comparison of Treatments for Frozen Shoulder: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Dec 1;3(12):e2029581. doi: 10.1001/jamanetworkopen.2020.29581. PMID 33326025
- [Background] Page MJ, Green S, Kramer S, Johnston RV, McBain B, Buchbinder R. Electrotherapy modalities for adhesive capsulitis (frozen shoulder). Cochrane Database Syst Rev. 2014 Oct 1;2014(10):CD011324. doi: 10.1002/14651858.CD011324. PMID 25271097
- [Background] Casarino V, Ciatti P, Martini A. Weighted spectral cluster bounds and a sharp multiplier theorem for ultraspherical Grushin operators. International Mathematics Research Notices. 2022;2022(12):9209-9274. doi:10.1093/imrn/rnab007
- [Background] Kelley MJ, Shaffer MA, Kuhn JE, Michener LA, Seitz AL, Uhl TL, Godges JJ, McClure PW. Shoulder pain and mobility deficits: adhesive capsulitis. J Orthop Sports Phys Ther. 2013 May;43(5):A1-31. doi: 10.2519/jospt.2013.0302. Epub 2013 Apr 30. No abstract available. PMID 23636125
- [Background] Corbacho B, Brealey S, Keding A, Richardson G, Torgerson D, Hewitt C, McDaid C, Rangan A; UK FROST trial team. Cost-effectiveness of surgical treatments compared with early structured physiotherapy in secondary care for adults with primary frozen shoulder : an economic evaluation of the UK FROST trial. Bone Jt Open. 2021 Aug;2(8):685-695. doi: 10.1302/2633-1462.28.BJO-2021-0075.R1. PMID 34420365
- [Background] Kim DH, Kim YS, Kim BS, Sung DH, Song KS, Cho CH. Is frozen shoulder completely resolved at 2 years after the onset of disease? J Orthop Sci. 2020 Mar;25(2):224-228. doi: 10.1016/j.jos.2019.03.011. Epub 2019 Apr 2. PMID 30952550
- [Background] Page P, Labbe A. Adhesive capsulitis: use the evidence to integrate your interventions. N Am J Sports Phys Ther. 2010 Dec;5(4):266-73. PMID 21655385
- [Background] Le HV, Lee SJ, Nazarian A, Rodriguez EK. Adhesive capsulitis of the shoulder: review of pathophysiology and current clinical treatments. Shoulder Elbow. 2017 Apr;9(2):75-84. doi: 10.1177/1758573216676786. Epub 2016 Nov 7. PMID 28405218
- [Background] Cao W, Chen J, Pu J, Fan Y, Cao Y. Risk Factors for the Onset of Frozen Shoulder in Middle-Aged and Elderly Subjects Within 1 Year of Discharge From a Hospitalization That Involved Intravenous Infusion: A Prospective Cohort Study. Front Med (Lausanne). 2022 Jun 20;9:911532. doi: 10.3389/fmed.2022.911532. eCollection 2022. PMID 35795630
- [Background] Sun G, Li Q, Yin Y, Fu W, He K, Pen X. Risk factors and predictive models for frozen shoulder. Sci Rep. 2024 Jul 3;14(1):15261. doi: 10.1038/s41598-024-66360-y. PMID 38956312